CLINICAL TRIAL: NCT06644287
Title: The Value of 68Ga-grazytracer PET in Monitoring Responses to Immunotherapy of Advanced Soft Tissue Sarcomas
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Deputy director, Ruijin Hospital
Other Study IDs: RuijinH 2024-279
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: Advanced Soft Tissue Sarcomas
Keywords: 68Ga-grazytracer PET/CT; Immunotherapy; advanced soft tissue sarcomas

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnosis of advanced soft tissue sarcomas: Patients diagnosis of advanced soft tissue sarcomas require immunotherapy or combination immunotherapy after evaluation

SUMMARY:
This study aims to investigate the value of 68Ga-grazytracer in predicting the efficacy of immunotherapy for advanced soft tissue sarcomas.

DETAILED DESCRIPTION:
The investigators will number all participants, create a medical record file, and record their basic information (gender, age) as well as contact information and medical history information. All participants will undergo a 68Ga-grazytracer PET/CT after 3 cycles of immunotherapy to evaluate response. The imaging response measurements will be compared with the histopathological or clinical assessment results as gold standard.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological and clinical diagnosis of advanced soft tissue sarcomas, pathological types include: fibrosarcoma, liposarcoma, undifferentiated pleomorphic sarcoma, epithelioid sarcoma, rhabdomyosarcoma, synovial sarcoma, alveolar soft-part sarcoma, leiomyosarcoma, clear cell sarcoma, malignant schwannoma, angiosarcoma.
2. Consider immunotherapy or combined immunotherapy based on clinical judgement.
3. Signed and dated informed consent form.
4. Commitment to comply with research procedures and co-operation in the implementation of the full research process.
5. Aged 6-80 years old.

Exclusion Criteria:

1. Patients with serious illnesses that researchers consider unsuitable for participation in this clinical study. Such as severe heart and lung failure, severe bone marrow suppression, severe liver and kidney dysfunction, etc.
2. Intestinal perforation, complete intestinal obstruction
3. Pregnant women and women who may be pregnant, women who are breastfeeding.
4. Non-compliant person

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients and outpatients at Ruijin Hospital who meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation the responses to immunotherapy of advanced soft tissue sarcomas | up to about 10 weeks
  The value of 68Ga-grazytracer PET in monitoring responses to immunotherapy of advanced soft tissue sarcomas
Standardized uptake value(SUV) | up to about 10 weeks
  SUV of 68Ga-grazytracer uptake on PET/CT images for tumor lesions
Target-to-background ratio(TBR) | up to about 10 weeks
  68Ga-grazytracer uptake ratio of tumor lesions to mediastinum and liver blood pool on PET/CT images.

SECONDARY OUTCOMES:
Progress free survival | 1 years
  Progress free survival
Overall survival | 1 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No